CLINICAL TRIAL: NCT02400450
Title: Assessment of Designer Functional Foods on Parameters of Metabolic and Vascular Status in Individuals With Prediabetes.
Brief Title: Designer Functional Foods on Parameters of Metabolic and Vascular in Prediabetes
Acronym: PREFFER-2014
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Science and Technology International Collaboration Fund (Unknown); Manitoba Agri-Health Research Network (Other)
Responsible Party: Principal Investigator, Dr. Carla Taylor, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B2014:041
Record Dates: First submitted 2015-02-11; First posted 2015-03-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pre-Diabetes
Keywords: Pre-diabetes; prediabetes; glycated hemoglobin; hemoglobin A1c; LDL cholesterol; Cholesterol; metabolic function; vascular function; functional food
MeSH Terms: conditions — Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functional Ingredient Group (Experimental): Participants will be provided with a mix of 6 study products to use over the 12 week trial (2 per day). These will be a) oatmeal, b) pancake mix, c) chocolate crunch bar, d) cranberry nut bar, e) anytime sprinkle, and f) smoothie mix. The food items will contain a standardized amount of functional ingredients.
  Interventions: Dietary Supplement: Functional Ingredient Group
- Control Ingredient Group (Placebo Comparator): The control group will receive a comparable set of food items that contain an equivalent amount of calories per portion but without the added functional ingredients.
  Interventions: Dietary Supplement: Control Ingredient Group

INTERVENTIONS:
Dietary Supplement: Functional Ingredient Group — Participants will be provided with a mix of 6 study products to use over the 12 week trial (2 per day). These will be a) oatmeal, b) pancake mix, c) chocolate crunch bar, d) cranberry nut bar, e) anytime sprinkle, and f) smoothie mix, standardized for the content of functional ingredients.
  Other Names: Step One Foods (TruHealthMD)
  Arms: Functional Ingredient Group
Dietary Supplement: Control Ingredient Group — The control group will receive a comparable set of food items to use over the 12 week trial (2 per day). These food items will contain an equivalent amount of calories per portion but without the additional functional ingredients.
  Arms: Control Ingredient Group

SUMMARY:
This is a multi-site, double-blind, randomized, controlled food intervention study being conducted at the Canadian Centre for Agri-Food Research in Health and Medicine (CCARM) in Winnipeg and the Mayo Clinic, Rochester, MN, to examine the effects of a portfolio of functional foods on blood glucose and lipids, and blood vessel function in individuals with prediabetes.

A total of 116 participants (n=58/site) with prediabetes (hemoglobin A1c ≥6.0 & <7.0 and no glucose-lowering medications) and body-mass index (BMI) 18-40 will be recruited for a 12-week clinical trial to determine the effect of eating 2 items containing functional ingredients daily compared to 2 similar items lacking the functional ingredients. Study foods provided are to be incorporated into participant's usual diet.

DETAILED DESCRIPTION:
This study will investigate the effect of a 12 week intervention with a portfolio of 7 food products and 7 comparator products for their effect on glycated hemoglobin, blood lipids, blood vessel function and metabolic parameters in persons with prediabetes. Prediabetes precedes the manifestation of type 2 diabetes and is therefore an appropriate target for dietary interventions. It is also associated with increased cardiovascular disease (CVD) risk because of the presence of abdominal obesity, elevated LDL-cholesterol and reduced vascular function. CVD risk will be assessed based on the profile of lipids and other factors in the blood as well using specialized equipment for non-invasive monitoring of blood vessel function.

If the foods prove beneficial for managing blood glucose levels, the publication of results in scientific journals and in lay documents will increase awareness and provide important information of the health benefits of these products for consumers, health professionals and the food industry. It will also help individuals who may be able to manage their illnesses in a healthful non-pharmaceutical nutritional approach and who may benefit from physician-prescribed nutritional counseling with a focus on foods known to improve certain disease biomarkers. At this time these approaches lack practicality and direct application to individuals who are interested in adopting a new dietary regime capable of disease prevention.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be eligible for participation in the study:

1. Male, or non-pregnant, non-lactating females, aged 21 - 75 years;
2. Glycated hemoglobin A1c ≥6.0% and <7.0%;
3. Body-mass index 18-40;
4. Able to read, write and communicate orally in English;
5. Willing to maintain a stable level of activity during participation in the study;
6. Willing to comply with protocol requirements and procedures;
7. Willing to provide written informed consent.

Exclusion Criteria:

Failure to meet any one of the above eligibility criteria will result in an inability to participate in the study. Participants will also be excluded if they have or require any of the following:

1 Previous diagnosis of diabetes or taking diabetes medications (glucose-lowering medications, insulin);

2. Previous diagnosis of cardiovascular disease (e.g. heart attack, stroke, peripheral artery disease), or taking lipid-lowering medications, or having a surgical procedure/intervention to treat cardiovascular disease (e.g. bypass surgery, stent). [Note that individuals with hypertension and/or taking anti-hypertensive medication are eligible to participate.];

3. Fasting LDL-cholesterol >160 mg/dL (>4.1 mmol/L);

4. Fasting triglycerides >400 mg/dL (>4.5 mmol/L);

5. Serum alanine aminotransferase (ALT) outside the normal range of 7-56 units/L;

6. Serum creatinine outside the normal range of 0.7-1.3 mg/dL for males and 0.6-1.1 mg/dL for females;

7. Conditions which affect normal nutrient absorption (e.g. Celiac disease, inflammatory bowel disease);

8. Untreated endocrine disorders with the potential to affect glucose and lipid metabolism;

9. In the previous 3 months and during the study, consumption of supplements or herbals in amounts that lower blood glucose or blood lipids (e.g. chromium, margarine with plant sterols, high fibre supplements such as Metamucil, cinnamon extract, ginseng, bitter melon, gamma-linolenic acid);

10. Food allergies or intolerances which severely limit the variety of study food products that can be consumed;

11. Eating philosophies or eating patterns that would limit or not include consumption of the study foods;

12. Any acute medical condition or surgical intervention within the past 3 months;

13. Conditions or medications which are likely to increase the risk to the participants or study personnel, or to reduce the ability of the participant to comply with the protocol, or affect the results;

14. Currently participating in or having participated in a food intervention study within the last month;

15. Inability to adhere to the study protocol;

16. Unable to obtain blood sample at the screening and/or baseline visit.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin (A1c) | 12 Weeks
  Assessments of glycated hemoglobin will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
LDL-Cholesterol | 12 Weeks
  Assessments of LDL-Cholesterol will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.

SECONDARY OUTCOMES:
Blood Lipids (Total Cholesterol, HDL-Cholesterol, and Triglycerides) | 12 Weeks
  Assessment of blood lipid profile will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
Blood Glucose | 12 Weeks
  Assessment of glucose will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
Insulin | 12 Weeks
  Assessment of insulin (and calculation of insulin sensitivity using HOMA-IR, QUICKI) will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
C-Reactive Protein | 12 Weeks
  Assessment of C-Reactive Protein will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
Advanced Glycation End-products (AGE) | 12 Weeks
  Assessment of advanced glycated endproducts (AGEs) using a non-invasive skin fluorescence device (AGE Reader from Diagnotipics Inc.) will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
Pulse Wave Analysis/Velocity (Blood Vessel Function) | 12 Weeks
  Assessment of blood vessel function (arterial compliance) via pulse-wave analysis and pulse wave velocity will be performed at the Baseline Visit (Day 1), Week 6 (Day 56) and Week 12 (Day 84) visits.
Biomarkers of Vascular Function | 12 Weeks
  Assessment of biomarkers of vascular function in acquired blood samples will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
Biomarkers of Inflammation, Oxidative Stress, Immune Function and Metabolism | Week 12
  Assessment of inflammation, oxidative stress, immune function and metabolism from acquired blood samples will be completed at Baseline Visit (Day 1), Week 6 (Day 42) and Week 12 visits (Day 84) visits.
Changes in composite measure of Anthropometrics | 12 Weeks
  Changes in anthropometrics, specifically weight, body mass index, waist and hip circumference will be compared to the Baseline Visit (Day 1) and will be acquired at the Week 6 (Day 56) and Week 12 (Day 84) visits. Changes in body fat composition as assessed via dual-energy x-ray absorptiometry (DEXA)) will be assesed at the Baseline Visit (Day 1) and Week 12 (Day 84) visit.
Blood Pressure | 12 Weeks
  Blood pressure will be measure and assessed for changes at the Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) visit.
Food Consumption Patterns | 12 Weeks
  Food consumption patterns will be assessed from Baseline Visit (Day 1) to Week 12 (Day 84) using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Lindstrom J, Louheranta A, Mannelin M, Rastas M, Salminen V, Eriksson J, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. The Finnish Diabetes Prevention Study (DPS): Lifestyle intervention and 3-year results on diet and physical activity. Diabetes Care. 2003 Dec;26(12):3230-6. doi: 10.2337/diacare.26.12.3230. PMID 14633807
- [Background] Diabetes Prevention Program Research Group; Knowler WC, Fowler SE, Hamman RF, Christophi CA, Hoffman HJ, Brenneman AT, Brown-Friday JO, Goldberg R, Venditti E, Nathan DM. 10-year follow-up of diabetes incidence and weight loss in the Diabetes Prevention Program Outcomes Study. Lancet. 2009 Nov 14;374(9702):1677-86. doi: 10.1016/S0140-6736(09)61457-4. Epub 2009 Oct 29. PMID 19878986
- [Background] Silva FM, Kramer CK, de Almeida JC, Steemburgo T, Gross JL, Azevedo MJ. Fiber intake and glycemic control in patients with type 2 diabetes mellitus: a systematic review with meta-analysis of randomized controlled trials. Nutr Rev. 2013 Dec;71(12):790-801. doi: 10.1111/nure.12076. Epub 2013 Nov 1. PMID 24180564
- [Background] Hlebowicz J, Drake I, Gullberg B, Sonestedt E, Wallstrom P, Persson M, Nilsson J, Hedblad B, Wirfalt E. A high diet quality is associated with lower incidence of cardiovascular events in the Malmo diet and cancer cohort. PLoS One. 2013 Aug 5;8(8):e71095. doi: 10.1371/journal.pone.0071095. Print 2013. PMID 23940694
- [Background] Deng R. A review of the hypoglycemic effects of five commonly used herbal food supplements. Recent Pat Food Nutr Agric. 2012 Apr 1;4(1):50-60. doi: 10.2174/2212798411204010050. PMID 22329631
- [Background] Lee T, Dugoua JJ. Nutritional supplements and their effect on glucose control. Adv Exp Med Biol. 2012;771:381-95. doi: 10.1007/978-1-4614-5441-0_27. PMID 23393691
- [Background] Shane-McWhorter L. Dietary supplements and probiotics for diabetes. Am J Nurs. 2012 Jul;112(7):47-53. doi: 10.1097/01.NAJ.0000415961.92674.d4. PMID 22739611
- [Background] Suksomboon N, Poolsup N, Boonkaew S, Suthisisang CC. Meta-analysis of the effect of herbal supplement on glycemic control in type 2 diabetes. J Ethnopharmacol. 2011 Oct 11;137(3):1328-33. doi: 10.1016/j.jep.2011.07.059. Epub 2011 Aug 5. PMID 21843614
- [Background] Perera PK, Li Y. Functional herbal food ingredients used in type 2 diabetes mellitus. Pharmacogn Rev. 2012 Jan;6(11):37-45. doi: 10.4103/0973-7847.95863. PMID 22654403
- [Background] Thondre PS. Food-based ingredients to modulate blood glucose. Adv Food Nutr Res. 2013;70:181-227. doi: 10.1016/B978-0-12-416555-7.00005-9. PMID 23722097
- [Background] Cheng DM, Kuhn P, Poulev A, Rojo LE, Lila MA, Raskin I. In vivo and in vitro antidiabetic effects of aqueous cinnamon extract and cinnamon polyphenol-enhanced food matrix. Food Chem. 2012 Dec 15;135(4):2994-3002. doi: 10.1016/j.foodchem.2012.06.117. Epub 2012 Jul 14. PMID 22980902
- [Background] Pawar K, Thompkinson DK. Multiple functional ingredient approach in formulating dietary supplement for management of diabetes: a review. Crit Rev Food Sci Nutr. 2014;54(7):957-73. doi: 10.1080/10408398.2011.621039. PMID 24499073
- [Background] Vinik AI. A medicinal food provides food for thought in managing diabetic neuropathy. Am J Med. 2013 Feb;126(2):95-6. doi: 10.1016/j.amjmed.2012.08.008. No abstract available. PMID 23331432
- [Background] Stringer DM, Taylor CG, Appah P, Blewett H, Zahradka P. Consumption of buckwheat modulates the post-prandial response of selected gastrointestinal satiety hormones in individuals with type 2 diabetes mellitus. Metabolism. 2013 Jul;62(7):1021-31. doi: 10.1016/j.metabol.2013.01.021. Epub 2013 Feb 26. PMID 23485142
- [Background] Welch RW, Antoine JM, Berta JL, Bub A, de Vries J, Guarner F, Hasselwander O, Hendriks H, Jakel M, Koletzko BV, Patterson CC, Richelle M, Skarp M, Theis S, Vidry S, Woodside JV; International Life Sciences Institute Europe Functional Foods Task Force. Guidelines for the design, conduct and reporting of human intervention studies to evaluate the health benefits of foods. Br J Nutr. 2011 Nov;106 Suppl 2:S3-15. doi: 10.1017/S0007114511003606. PMID 22129662
- [Background] Jenkins DJ, Kendall CW, Banach MS, Srichaikul K, Vidgen E, Mitchell S, Parker T, Nishi S, Bashyam B, de Souza R, Ireland C, Josse RG. Nuts as a replacement for carbohydrates in the diabetic diet. Diabetes Care. 2011 Aug;34(8):1706-11. doi: 10.2337/dc11-0338. Epub 2011 Jun 29. PMID 21715526 (Retraction: PMID 26798151 Diabetes Care. 2016 Feb;39(2):319)
- See also: Canadian Centre for Agri-Food Research in Health and Medicine — http://www.ccarm.ca